CLINICAL TRIAL: NCT00874055
Title: The Presence of Friends Increases Food Intake in Youth
Status: Completed | Type: Observational
Sponsor: University at Buffalo (Other)
Responsible Party: Sarah-Jeanne Salvy, Ph.D., University at Buffalo, Division of Behavioral Medicine
Other Study IDs: DB2213; 1R01HD057190-01A1 (NIH)
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2009-04-02 (Estimated); Status verified 2009-04

CONDITIONS: Total Caloric Intake; Nutrient Dense Caloric Intake; Energy Dense Caloric Intake
Keywords: social influence; friends; eating behavior; childhood overweight
MeSH Terms: conditions — Feeding Behavior; Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
Participants will be matched with either their friend or an unfamiliar peer who is the same gender and about the same age. Participants will have 45 minutes of free-play in an experimental room where they will have free access to energy-dense and nutrient-dense foods and an assortment of games and puzzles.

The investigators predict that participants eating with a friend will eat significantly more than participants eating with an unfamiliar peer. The investigators also predict that overweight participants eating with an overweight partner will eat significantly more than participants eating with a non overweight participant.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls ages 9-15
* Between 15th and 95th BMI percentile for their age

Exclusion Criteria:

* Sickness, psychopathology or developmental disabilities
* Participant has a cold or upper respiratory distress
* Food allergies to the study food
* Participant is on medication or has a medical condition that could influence taste, appetite or olfactory sensory responsiveness.

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Boys and girls between the ages of 9-15.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2007-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah J Salvy, Ph.D., Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Division of Behavioral Medicine, Buffalo, New York, United States

REFERENCES:
- [Derived] Salvy SJ, Howard M, Read M, Mele E. The presence of friends increases food intake in youth. Am J Clin Nutr. 2009 Aug;90(2):282-7. doi: 10.3945/ajcn.2009.27658. Epub 2009 Jun 17. PMID 19535431